CLINICAL TRIAL: NCT07021157
Title: A Randomized, Double-blind, Placebo-controlled, Phase I Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetic Characteristics of Single-dose Increasing of SK-08 Tablets in Healthy Participants
Brief Title: A Study to Evaluate the Safety, Tolerability and PK of SK-08
Acronym: SK-08
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Consun Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-CP-SK08-01
Record Dates: First submitted 2025-05-12; First posted 2025-06-13 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-05

CONDITIONS: Chronic Kidney Disease(CKD)
Keywords: Chronic Kidney Disease(CKD)
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SK-08 (Experimental): Seven sequential dose groups（A1-A7） will be evaluated: 5 mg, 7.5mg,12.5 mg, 20 mg, 30 mg, 45 mg, and 60 mg.
  SK-08 were given once for 5mg, 7.5mg,12.5 mg, 30 mg, 45 mg, and 60 mg dose groups.
  Interventions: Drug: SK-08
- Placebo (Placebo Comparator): Seven sequential dose groups（A1-A7） will be evaluated: 5 mg, 7.5mg,12.5 mg, 30 mg, 45 mg, and 60 mg.
  Placebo were given once for 5mg, 7.5mg,12.5 mg, 30 mg, 45 mg, and 60 mg dose groups.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SK-08 — Dose groups of 5 mg, 7.5mg,12.5 mg, 30 mg, 45 mg, and 60 mg were given SK-08 once.
  Arms: SK-08
Drug: Placebo — Dose groups of 5 mg, 7.5mg,12.5 mg, 30 mg, 45 mg, and 60 mg were given placebo once.
  Arms: Placebo

SUMMARY:
The trial is conducted in a single-center, randomized, double-blind, placebo-controlled, dose-increasing design. To evaluate the safety, tolerability, pharmacokinetics(PK) ,and pharmacodynamics (PD) characteristics of SK-08 in healthy participants.

DETAILED DESCRIPTION:
The trial is conducted in a single-center, randomized, double-blind, placebo-controlled, dose-increasing design. To evaluate the safety, tolerability, pharmacokinetics(PK) ,and pharmacodynamics (PD) characteristics of SK-08 in healthy participants. Seven dose groups (A1 to A7) were preset. A total of 48 healthy subjects were planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female participants aged 18 to 45 years (inclusive).
2. Male participants: Body weight ≥50 kg; Female participants: Body weight ≥45 kg; Body mass index (BMI) between 19.0 and 26 kg/m².
3. Participants must have no plans for conception during the trial and for 3 months after the last dose, and must voluntarily use effective contraception with no plans for sperm or egg donation .
4. Capable of understanding and voluntarily providing written informed consent prior to any study-related procedures.

Exclusion Criteria:

1. Have a specific history of allergies or have an allergic constitution；
2. Have a history of chronic diseases or severe diseases in the cardiovascular, liver, kidney, biliary tract, respiratory, blood and lymphatic, endocrine, immune, mental, neuromuscular, gastrointestinal systems, etc.
3. Developed acute diseases from 2 weeks before screening to before randomization ;
4. Patients with previous or current hypotension or insufficient blood volume, intracranial hypertension or cerebral hemorrhage, or those with ocular diseases (such as angle-closure glaucoma), who are not suitable for inclusion after assessment by the researcher;
5. Those with clinical significance hypokalemia, hyperkalemia, hypomagnesemia, hypermagnesemia, hypocalcemia, and hypercalcemia;
6. Those who have used any drugs or health supplements from 2 weeks before screening to randomization ;
7. Any drugs that may interact with this product have been used from 30 days before screening to randomization, such as CYP450 inhibitors or inducers ;
8. Those who have undergone major surgical operations from 6 months before screening , or who plan to undergo surgery during the study period, or who have undergone surgeries as judged by the investigator to affect drug absorption, distribution, metabolism, and excretion;
9. Those who have received live attenuated vaccine inoculation from 2 weeks before screening to randomization or those who need to receive live attenuated vaccine inoculation during the trial;
10. Those who had a history of alcohol abuse within one year before screening；
11. Those who smoked more than 5 cigarettes per day on average within 3 months before screening and before randomization, or were unable to stop using any tobacco products during the trial period;
12. Those who cannot tolerate venipuncture/indwelling needles or have a history of fainting from needles or blood ;
13. Other researchers determined that the subjects were not suitable to participate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-03-09 (Actual); Primary Completion 2025-08-07 (Estimated); Study Completion 2025-08-07 (Estimated)

PRIMARY OUTCOMES:
Safety Evaluation | up to Day 12
  The occurrence of AE during the experiment

SECONDARY OUTCOMES:
PK Evaluation（Cmax） | within 1 hour pre-dosing and at 0.5 hour, 1 hour, 1.5 hour, 2 hour, 2.25hour，2.5 hour, 2.75hour，3 hour, 3.5hour，4 hour, 5hour，6 hour, 8 hour, 12 hour, 24 hour , 48 hour, 72 hour and 96hour post-dosing
  Pharmacokinetic characteristics after administration (Cmax）
PK Evaluation（Tmax） | within 1 hour pre-dosing and at 0.5 hour, 1 hour, 1.5 hour, 2 hour, 2.25hour，2.5 hour, 2.75hour，3 hour, 3.5hour，4 hour, 5hour，6 hour, 8 hour, 12 hour, 24 hour , 48 hour, 72 hour and 96hour post-dosing
  Pharmacokinetic characteristics after administration
PK Evaluation（ AUC0-T） | within 1 hour pre-dosing and at 0.5 hour, 1 hour, 1.5 hour, 2 hour, 2.25hour，2.5 hour, 2.75hour，3 hour, 3.5hour，4 hour, 5hour，6 hour, 8 hour, 12 hour, 24 hour , 48 hour, 72 hour and 96hour post-dosing
  Pharmacokinetic characteristics after administration (AUC0-T）
PK Evaluation ( AUC0-∞） | within 1 hour pre-dosing and at 0.5 hour, 1 hour, 1.5 hour, 2 hour, 2.25hour，2.5 hour, 2.75hour，3 hour, 3.5hour，4 hour, 5hour，6 hour, 8 hour, 12 hour, 24 hour , 48 hour, 72 hour and 96hour post-dosing
  Pharmacokinetic characteristics after administration ( AUC0-∞）
PD Evaluation（Heart rate） | within 1.0hour pre-dosing, and at 1.0hour, 2.0hour, 4.0hour, 6.0h, and 12.0h post dosing
  Heart rate
PD Evaluation（blood pressure） | within 1.0hour pre-dosing, and at 1.0hour, 2.0hour, 4.0hour, 6.0h, and 12.0h post dosing
  blood pressure
PD Evaluation（changes in cGMP concentration levels） | within 1.00 hour pre-dosing and 0.50 hour, 1hour,1.5hour,2hour,2.5hour,3hour,4hour,5hour,6hour,8hour,12hour post-dosing
  changes in cGMP concentration levels
QT interval analysis indicators（QTcF） | With in1hour pre-dosing,and at 0.5hour、1.0hour、1.5hour、2.0hour、4.0hour、6.0hour、12.0hour、24.0hour post-dosing
  QTcF
QT interval analysis indicators（ΔQTcF） | With in1hour pre-dosing,and at 0.5hour、1.0hour、1.5hour、2.0hour、4.0hour、6.0hour、12.0hour、24.0hour post-dosing
  ΔQTcF

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital，Zhejiang University, Hangzhou, Zhejiang, China